CLINICAL TRIAL: NCT05329311
Title: The Effect of Enhanced Recovery After Thoracic Surgery Protocol on Inflammatory Markers
Brief Title: Enhanced Recovery After Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2319
Record Dates: First submitted 2022-03-16; First posted 2022-04-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Enhanced Recovery After Thoracic Surgery Protocol; C-reactive Protein; White Blood Cell Count; Neutrophil/Lymphocyte Ratio; Plathelet/ Lymphocyte Ratio; Lymphocyte/Monocytes Ratio; Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERATS protocol applied: Inflammatory parameters of the operated patients by applying the ERATS protocol will be investigated.
  Interventions: Procedure: ERATS protocol applied
- ERATS protocol not applied: Inflammatory parameters of patients who were operated without the ERATS protocol will be investigated.
  Interventions: Procedure: ERATS protocol not applied

INTERVENTIONS:
Procedure: ERATS protocol applied — Inflammatory parameters (such as; C-reactive protein (CRP), white blood cell count, neutrophil/lymphocyte ratio (NLR), platelet/ lymphocyte ratio (PLR), lymphocyte/monocytes ratio (LMR) of the operated patients by applying the ERATS protocol will be investigated.
  Groups: ERATS protocol applied
Procedure: ERATS protocol not applied — Inflammatory parameters (such as; C-reactive protein (CRP), white blood cell count, neutrophil/lymphocyte ratio (NLR), platelet/ lymphocyte ratio (PLR), lymphocyte/monocytes ratio (LMR) of the operated patients by applying without the ERATS protocol will be investigated.
  Groups: ERATS protocol not applied

SUMMARY:
Despite significant advances in perioperative care, major complications continue to be seen in patients undergoing major surgery. Enhanced recovery after surgery (ERAS) protocols are perioperative care practices designed to reduce perioperative complications, maintain preoperative organ function, and provide early recovery by reducing the psychological and physiological response to major surgery and the intense stress response that develops following surgery. In this context, ERAS protocols have been established for many surgical procedures. One is the thoracic ERAS (ERATS) protocol applied to thoracic surgery, and the evidence for ERATS is increasing; literature data support the application of ERATS. However, there are limited studies on the application of ERAS protocols to thoracic surgery, and more studies are needed to develop ERATS protocols.

Postoperative complications may be reduced in patients who are treated with the ERAS protocol, their length of hospital stay (LOS) may be shortened, and patients may regain their initial functions faster. Objectively, a marker indicating whether the ERAS protocol can be implemented effectively has not yet been demonstrated. Reducing postoperative inflammation is thought to reduce LOS. Based on this, the investigators think that the early recovery seen in patients who undergo ERAS is due to the effect of ERAS protocols on the inflammatory process. Therefore, laboratory parameters such as C-reactive protein (CRP), white blood cell count, neutrophil/lymphocyte ratio (NLR), platelet/lymphocyte ratio (PLR), lymphocyte/monocytes ratio (LMR) may differ in patients who have undergone the ERAS protocol compared to patients who have not. These parameters have been evaluated comprehensively in studies as inflammatory parameters. In addition, clinical studies indicate that the C-reactive protein to albumin ratio (CAR) can be used as inflammatory and prognostic markers. Also, the investigators hypothesized that inflammatory parameters used in routine clinical follow-up may be effective in evaluating the clinical consequences of ERATS protocols. In this study, the investigators aimed to evaluate the effects of the ERATS protocol on postoperative inflammatory parameters and investigate whether these parameters have a role in evaluating the effectiveness of the ERATS protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-80 years of
* Patients underwent elective thoracic surgery,
* American Society of Anesthesiologists (ASA) I-II-III
* Body mass index (BMI) between 18.5-35 kg/m2

Exclusion Criteria:

* Patients with systemic inflammatory diseases
* Patients with a history of anti-inflammatory and anti-allergic drugs,
* Patients with a history of corticosteroid usage,
* Patients who had received intraoperative blood product transfusions,
* Patients who had previously undergone thoracic surgery,
* Patients with missing data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients between 18-80 years of age who had undergone elective thoracic surgery, whose physical condition was I-II-III according to the ASA, and whose BMI was between 18.5-35 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Postoperative C-reactive protein | Change from baseline CRP on the first, third, and fifth postoperative days
  The postoperative C-reactive protein (CRP) (mg/L) of patients who had thoracic surgery will be investigated from the hospital archive.
  The results of the patients who were operated on according to the ERATS protocol and who were operated on without ERATS protocol did will be compared.
Postoperative white blood cell count | Change from baseline WBC on the first, third, and fifth postoperative days
  The postoperative white blood cell count (WBC) (x10^3/µL) of patients who had thoracic surgery will be investigated from the hospital archive.
  The results of the patients who were operated on according to the ERATS protocol and who were operated on without ERATS protocol did will be compared.
Postoperative neutrophil/lymphocyte ratio | Change from baseline NLR on the first, third, and fifth postoperative days
  The postoperative neutrophil/lymphocyte ratio (NLR) of patients who had thoracic surgery will be investigated from the hospital archive.
  The results of the patients who were operated on according to the ERATS protocol and who were operated on without ERATS protocol did will be compared.
Postoperative platelet/lymphocyte ratio | Change from baseline PLR on the first, third, and fifth postoperative days
  The postoperative platelet/lymphocyte ratio (PLR) of patients who had thoracic surgery will be investigated from the hospital archive.
  The results of the patients who were operated on according to the ERATS protocol and who were operated on without ERATS protocol did will be compared.
Postoperative lymphocyte/monocytes ratio | Change from baseline LMR on the first, third, and fifth postoperative days
  The postoperative lymphocyte/monocytes ratio (LMR) of patients who had thoracic surgery will be investigated from the hospital archive.
  The results of the patients who were operated on according to the ERATS protocol and who were operated on without ERATS protocol did will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)